CLINICAL TRIAL: NCT00930930
Title: A Phase II Neo-Adjuvant Study of Cisplatin, Paclitaxel With or Without RAD001 in Patients With Triple-negative Locally Advanced Breast Cancer.
Brief Title: Cisplatin and Paclitaxel With or Without Everolimus in Treating Patients With Stage II or Stage III Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ingrid Mayer, MD, Assistant Professor of Medicine; Clinical Director, Breast Cancer Program; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VICC BRE 0904; P30CA068485 (NIH); VU-VICC-BRE-0904; IRB# 090291
Record Dates: First submitted 2009-07-01; First posted 2009-07-02 (Estimated); Results first posted 2015-05-07 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Breast Cancer
Keywords: triple-negative breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms; Breast Neoplasms, Male | interventions — Cisplatin; Everolimus; Paclitaxel; Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cisplatin and Paclitaxel + RAD001 (Experimental): Cisplatin 25 mg/m2 IV weekly + RAD001 5 mg PO daily for 1 week followed by Cisplatin 25 mg/m2 IV + Paclitaxel 80 mg/m2 IV weekly + RAD001 5 mg PO daily for 11 weeks
  Interventions: Drug: cisplatin; Drug: everolimus; Drug: paclitaxel; Procedure: Venous blood draw
- Cisplatin and Paclitaxel + Placebo (Active Comparator): Cisplatin 25 mg/m2 IV weekly + placebo PO daily for 1 week followed by Cisplatin 25 mg/m2 IV + Paclitaxel 80 mg/m2 IV weekly + placebo PO daily for 11 weeks
  Interventions: Drug: cisplatin; Drug: paclitaxel; Other: placebo; Procedure: Venous blood draw

INTERVENTIONS:
Drug: cisplatin — Given IV
Drug: everolimus — Given orally
  Arms: Cisplatin and Paclitaxel + RAD001
Drug: paclitaxel — Given IV
Other: placebo — Given orally
  Arms: Cisplatin and Paclitaxel + Placebo
Procedure: Venous blood draw — Venous blood (2-3 tablespoons) will be taken for germline DNA analysis to complement the correlative studies in the tumor tissue. Blood can be drawn at any time prior, during, or after completion of study treatment

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving chemotherapy together with everolimus before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. It is not yet known whether cisplatin and paclitaxel are more effective when given together with or without everolimus in treating patients with breast cancer.

PURPOSE: This randomized phase II trial is studying how well cisplatin and paclitaxel work when given together with or without everolimus in treating patients with stage II or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the pathological complete response in patients with triple-negative, stage II or III breast cancer treated with neoadjuvant cisplatin and paclitaxel with or without everolimus.

Secondary

* To determine the safety profile of these treatment regimens.
* To evaluate tumor response to these treatment regimens as measured by ultrasound before definitive surgery.
* To evaluate the rate of breast conservation surgery after treatment with these regimens.
* To determine treatment-mediated changes in cell cycle position, proliferation, and apoptosis as well as status, levels, and phosphorylation state of S6K, p53, p73, and p63 and select p53 family target genes before and after initiation of paclitaxel.
* To isolate RNA and generate microarray data sets from pre- and post-treatment biopsy material to identify a pre-treatment gene signature that will predict response.
* To isolate RNA and generate microarray data sets from pre- and post-treatment biopsy material to identify a change in gene signature after the first treatment that will predict response.
* To isolate RNA and generate microarray data sets from pre- and post-treatment biopsy material to determine if previously established p63 and p73 gene signatures predict response to treatment.
* To isolate RNA and generate microarray data sets from pre- and post-treatment biopsy material to determine if a change will be observed in p63 and p73 gene signatures between pre- and post-treatment biopsies.
* To isolate RNA and generate microarray data sets from pre- and post-treatment biopsy material to determine if triple-negative breast cancers can be clustered into different subtypes on the basis of gene expression, given the size of the microarray data set that will be generated from this clinical trial and previous clinical trials (> 100 tumors).
* To isolate RNA and generate microarray data sets from pre- and post-treatment biopsy material to determine if p63 and p73 gene signatures can sub-classify triple-negative breast cancers.

OUTLINE: This is a multicenter study. Patients are stratified according to initial lymph node status (positive vs negative involvement) and tumor grade (low or intermediate vs high). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive cisplatin IV over 1 hour and oral everolimus once weekly in weeks 1-12 and paclitaxel IV over 1 hour once weekly in weeks 4-12 in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive cisplatin IV over 1 hour and oral placebo once weekly in weeks 1-12 and paclitaxel IV over 1 hour once weekly in weeks 4-12 in the absence of disease progression or unacceptable toxicity.

Approximately 3-6 weeks after the completion of neoadjuvant therapy, patients undergo partial or total mastectomy with lymph node evaluation. Patients may then receive additional chemotherapy or radiotherapy.

Patients undergo ultrasound-guided core biopsies at baseline and in weeks 1, 4, and 12 for analysis of proliferation, apoptosis, and pathway activity markers via IHC or western blotting and RNA microarrays.

Patients are followed up within 3 weeks after surgery.

ELIGIBILITY:
Eligibility criteria

-Maximum number of patients will include two-thirds of the patients in Arm 1 and one-third of the patients for Arm 2 (total of 145 patients). Estimated time for accrual with ~ 3 patients/month would be ~ 3.5 years.

Inclusion criteria:

* Patients must provide informed written consent.
* Patient must be ≥ 18 years of age.
* ECOG performance status 0-1.
* Clinical stage II or stage III triple-negative (ER and/or PR no staining or weak staining in less than or equal to 10% cells by immunohistochemistry [IHC] and HER2-negative by Herceptest [0, 1+] or FISH) invasive mammary carcinoma, confirmed by histological analysis.
* Patients who have measurable* residual tumor at the primary site

  *Measurable disease: any mass that can be reproducibly measured by physical examination, mammogram, and/or ultrasound and can be accurately measured in at least one dimension (longest diameter to be recorded) as 10 mm (1 cm), either in the breast or axillary lymph nodes.
* Available core biopsies from the time of diagnosis. Fresh tissue must be obtainable at baseline or fresh tissue biopsy prior to treatment initiation.
* Patients who will undergo surgical treatment with either segmental resection or total mastectomy.
* Patients must have adequate hematologic, hepatic, and renal function. All tests must be obtained less than 4 weeks from study entry. This includes:
* ANC >/=1500/mm3
* Platelet count >/=100,000/mm3
* Creatinine </=1.5X upper limits of normal
* Bilirubin, SGOT, SGPT </=1.5X upper limits of normal*

  * for patients with Gilbert"s syndrome, direct bilirubin will be measured instead of total bilirubin.
* The patient must have not had anyprior chemotherapy for primary breast cancer.
* Patients with a prior history of contra-lateral breast cancer are eligible if they have no evidence of recurrence of their initial primary breast cancer within the last 5 years.
* Able to swallow and retain oral medication.
* Four days prior to biopsy procedures patients must be off medications that could increase risk of bleeding (i.e. ASA, NSAIDS, Coumadin, heparin products)
* Potential subjects must complete all screening assessments as outlined in the protocol.
* The pre-menopausal patient of childbearing potential must have had a negative pregnancy test and agreed to use birth control methods while participating in the study. Note: Women of childbearing potential and their male counterparts should use a barrier method of contraception during and for 3 months following protocol therapy.

Ineligibility Criteria

Exclusion Criteria:

* Locally recurrent breast cancer.
* Pregnant or lactating women.
* Evidence of distant metastatic disease (i.e. lung, liver, bone, brain, etc.)
* Use of CYP3A4 modifiers (Appendix A)
* Serious medical illness that in the judgment of the treating physician places the patient at high risk of operative mortality.
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel.
* History of other malignancy. Subjects who have been disease-free for 5 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinomas are eligible.
* History of hepatitis B or hepatitis C. If patient is judged to be at risk for having had exposure to viral B or C hepatitis (i.e. illicit IV drug use, blood transfusion prior to 1990, body piercing, tattoos, etc.), appropriate testing should be performed (i.e. Hepatitis B surface antigen antibody, and Hepatitis C antibody)
* Active or uncontrolled infection requiring parenteral antibiotics.
* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.
* Symptomatic neuropathy (≥ grade 2).
* Concurrent anti-cancer therapy (chemotherapy, radiation therapy, surgery, immunotherapy, hormonal therapy, or any other biologic therapy) other than the ones specified in the protocol.
* Concurrent treatment with an investigational agent.
* Used an investigational drug within 15 days or 5 half-lives, whichever is longer, preceding the first dose of randomized therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2009-06; Primary Completion 2013-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Mayer, M.D., Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (8):
- United States (8):
  - University of Alabama, Birmingham, Alabama
  - University of Mississippi Medical Center Research Institute, Jackson, Mississippi
  - Hershey Medical Center, Hershey, Pennsylvania
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - MBCCOP - Meharry Medical College - Nashville, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - The Methodist Hospital Research Institute, Houston, Texas
  - University of Virginia Health Sciences Center, Charlottesville, Virginia

REFERENCES:
- [Derived] Jovanovic B, Sheng Q, Seitz RS, Lawrence KD, Morris SW, Thomas LR, Hout DR, Schweitzer BL, Guo Y, Pietenpol JA, Lehmann BD. Comparison of triple-negative breast cancer molecular subtyping using RNA from matched fresh-frozen versus formalin-fixed paraffin-embedded tissue. BMC Cancer. 2017 Apr 4;17(1):241. doi: 10.1186/s12885-017-3237-1. PMID 28376728
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Vanderbilt-Ingram Cancer Center, multi-site intervention study included 7 additional cancer centers. It opened to enrollment in June 2009 and ran through May 2013.
Pre-assignment Details: One hundred forty-seven patients enrolled in this study. Two patients were not eligible to participate.
Groups:
- Arm I: Cisplatin 25 mg/m2 IV weekly + RAD001 5 mg PO daily for 1 week followed by Cisplatin 25 mg/m2 IV + Paclitaxel 80 mg/m2 IV weekly + RAD001 5 mg PO daily for 11 weeks
  cisplatin: Given IV
  everolimus: Given orally
  paclitaxel: Given IV
  Venous blood draw: Venous blood (2-3 tablespoons) will be taken for germline DNA analysis to complement the correlative studies in the tumor tissue. Blood can be drawn at any time prior, during, or after completion of study treatment
- Arm II: Cisplatin 25 mg/m2 IV weekly + placebo PO daily for 1 week followed by Cisplatin 25 mg/m2 IV + Paclitaxel 80 mg/m2 IV weekly + placebo PO daily for 11 weeks
  cisplatin: Given IV
  paclitaxel: Given IV
  placebo: Given orally
  Venous blood draw: Venous blood (2-3 tablespoons) will be taken for germline DNA analysis to complement the correlative studies in the tumor tissue. Blood can be drawn at any time prior, during, or after completion of study treatment
Period: Overall Study
Arm/Group | Arm I | Arm II
Started | 96 | 49
Completed | 75 | 40
Not Completed | 21 | 9
Not completed — Death | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Adverse Event | 13 | 3
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Disease progression | 2 | 3
Not completed — excessive lapse btw txs, not eligible | 0 | 1
Not completed — patients not compliant | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I | Arm II | Total
Number analyzed (Participants) | 96 | 49 | 145
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 52 [42.8 to 57.2] | 52 [43 to 58] | 52 [43 to 58]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 87 | 46 | 133
  >=65 years | 9 | 3 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 49 | 145
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 96 | 49 | 145

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Pathological Complete Response
Description: Pathological complete response is defined as no residual tumor on histopathological analysis of both breast and axillary contents.
Time Frame: at time of surgery, week 15-18
Population: Number of patients that had complete response. Specimens containing only non-invasive disease will be classified as complete pathologic responders
Measure: Number; unit: participants
Arm/Group | Cisplatin and Paclitaxel + RAD001 | Cisplatin and Paclitaxel + Placebo
Number analyzed (Participants) | 88 | 44
participants | 34 | 17

2. Secondary Outcome: Number of Patients That Underwent Breast Conservation Surgery
Description: Defined as patients that did not undergo complete removal of a cancerous breast (mastectomy).
Time Frame: at the time of surgery, week 15-18
Population: participants that had breast conservation surgery
Measure: Number; unit: participants
Arm/Group | Cisplatin and Paclitaxel + RAD001 | Cisplatin and Paclitaxel + Placebo
Number analyzed (Participants) | 96 | 49
participants | 38 | 19

3. Secondary Outcome: Clinical Tumor Response to Neoadjuvant Therapy as Measured by Ultrasound Immediately Before Surgery
Description: Per RECIST criteria v. 1.0: measurable lesions: complete response (CR) disappearance of target lesions, partial response (PR) > 30% decrease in the sum of the longest diameter (LD) of target lesions, progressive disease (PD) > 20% increase in the sum of the LD of target lesions or appearance of new lesions, stable disease (SD) neither sufficient decrease nor increase of the sum of smallest sum of the LD of target lesions
Time Frame: After treatment, week 12-15
Population: Patients reported by best overall response data. Patients are excluded if best overall response data is not accessible or not evaluable.
Measure: Number; unit: participants
Arm/Group | Cisplatin and Paclitaxel + RAD001 | Cisplatin and Paclitaxel + Placebo
Number analyzed (Participants) | 96 | 48
participants
  Complete Response | 48 | 23
  Partial Response | 27 | 19
  Stable Disease | 18 | 5
  Progressive Disease | 2 | 0
  Not Evaluable | 1 | 1

4. Secondary Outcome: Number of Patients With Each Worst-grade Toxicity Response
Description: Tables represent the number of patients with their worst-grade toxicity at each of five grades (grade 1, least severe to grade 5, most severe) following NCI Common Toxicity Criteria. Not all participants necessarily have an adverse event, thus not everyone will be accounted for in worst-grade toxicities. Likewise, one participant can potentially have more than one event in various grades 1-5 which accounts for the difference in number of patients analyzed and total number in the worst-grade toxicity tables.
Time Frame: week 12
Population: Total number of patients reported with any toxicity related to study treatment.
Measure: Number; unit: participants
Arm/Group | Cisplatin and Paclitaxel + RAD001 | Cisplatin and Paclitaxel + Placebo
Number analyzed (Participants) | 96 | 49
participants
  Number of patients with worst-grade toxicity 1 | 9 | 5
  Number of patients with worst-grade toxicity 2 | 40 | 28
  Number of patients with worst-grade toxicity 3 | 39 | 9
  Number of patients with worst-grade toxicity 4 | 3 | 1
  Number of patients with worst-grade toxicity 5 | 0 | 0

5. Other Pre Specified Outcome: Therapy-mediated Changes in Cell Cycle Position, Proliferation, and Apoptosis as Well as Status, Levels, and Phosphorylation State of p53, p73, and p63 and Select p53 Family Target Genes
Description: To determine the relevance of pathway modulation in triple negative breast cancer cell networking
Time Frame: Before treatment, on day 3-5 of week 1, and at week 12
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Ability of p63 and p73 Gene Signatures to Predict Patient Response
Description: To determine the levels of P63 and p73 in order to correlate these levels with patient response to treatment to help define a biomarker signature associated with p63/p73 dependence in triple negative breast cancers
Time Frame: Before treatment, on day 3-5 of week 1, and at week 12
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year, 2 months
Arm/Group | Arm I | Arm II
Serious Adverse Events (participants affected / at risk) | 22/96 | 6/49
Other Adverse Events (participants affected / at risk) | 96/96 | 49/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=96) | Arm II (N=49)
Allergic reaction to study drug (Immune system disorders) | 1 (1) | 0 (0)
Dehydration (Gastrointestinal disorders) | 5 (5) | 1 (1)
hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
mental status altered (Psychiatric disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
cardiac ischemia/infarction (Cardiac disorders) | 1 (1) | 0 (0)
cerebrovascular ischemia (Vascular disorders) | 0 (0) | 1 (1)
colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
creatinine increased (Investigations) | 3 (3) | 0 (0)
diarrhea (Gastrointestinal disorders) | 5 (5) | 0 (0)
dizziness (Nervous system disorders) | 1 (1) | 0 (0)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
edema (General disorders) | 1 (1) | 0 (0)
fatigue (General disorders) | 2 (2) | 0 (0)
Fever with absence of neutropenia (General disorders) | 5 (5) | 0 (0)
flu-like symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
hemaglobin increased (Investigations) | 2 (2) | 0 (0)
infection- respiratory (Infections and infestations) | 5 (5) | 1 (1)
infection with unknown ANC (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Seroma (Infections and infestations) | 0 (0) | 1 (1)
infection - other (Infections and infestations) | 0 (0) | 1 (1)
ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
pain - chest (General disorders) | 1 (1) | 0 (0)
pain - extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
sinus tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
syncope (Vascular disorders) | 2 (2) | 2 (2)
Thrombosis (Vascular disorders) | 3 (3) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
distal small bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=96) | Arm II (N=49)
Alkaline Phosphatase (Metabolism and nutrition disorders) | 14 (21) | 4 (5)
Allergic reaction - including drug fever (Immune system disorders) | 14 (14) | 3 (3)
allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 6 (6)
Allergy - other (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1)
Serum glutamic pyruvic transaminase (Metabolism and nutrition disorders) | 23 (33) | 5 (7)
Anorexia (Metabolism and nutrition disorders) | 7 (8) | 7 (7)
Arthritis (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3)
Serum glutamic oxaloacetic transaminase (Metabolism and nutrition disorders) | 30 (36) | 4 (5)
hypocalcemia (Metabolism and nutrition disorders) | 19 (27) | 7 (7)
Cardiac General (Cardiac disorders) | 10 (11) | 1 (1)
hypercholesteremia (Metabolism and nutrition disorders) | 6 (6) | 3 (3)
Constipation (Gastrointestinal disorders) | 35 (38) | 19 (20)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 20 (20) | 8 (8)
General Disorders, other (General disorders) | 9 (10) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (15) | 5 (5)
Rashes (Skin and subcutaneous tissue disorders) | 38 (41) | 16 (17)
Diarrhea (Gastrointestinal disorders) | 44 (49) | 13 (14)
Dizziness (Nervous system disorders) | 7 (7) | 7 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 7 (8)
Edema (Renal and urinary disorders) | 14 (23) | 4 (4)
fatigue (General disorders) | 69 (83) | 36 (44)
Flushing (Vascular disorders) | 6 (6) | 15 (15)
Abdominal cramping (Gastrointestinal disorders) | 5 (5) | 6 (7)
Heartburn, dyspepsia, reflux, GERD (Gastrointestinal disorders) | 47 (48) | 20 (20)
Mucositis oral (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 0 (0)
hyperglycemia (Metabolism and nutrition disorders) | 45 (56) | 18 (27)
hypoglycemia (Metabolism and nutrition disorders) | 4 (4) | 3 (5)
alopecia (Skin and subcutaneous tissue disorders) | 32 (33) | 11 (11)
Hypertension (Vascular disorders) | 24 (24) | 15 (15)
infection - lung (Infections and infestations) | 5 (5) | 0 (0)
Infection - sinus (Infections and infestations) | 6 (6) | 2 (2)
Infection - Other (Infections and infestations) | 6 (6) | 5 (5)
infection - urinary (Renal and urinary disorders) | 7 (7) | 1 (1)
Insomnia (Psychiatric disorders) | 20 (20) | 10 (10)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 66 (104) | 32 (33)
Lymphopenia (Blood and lymphatic system disorders) | 7 (8) | 2 (2)
hypermagnesemia (Metabolism and nutrition disorders) | 11 (11) | 7 (7)
Metabolic/laboratory - other (Metabolism and nutrition disorders) | 23 (25) | 13 (13)
anxiety (Psychiatric disorders) | 28 (28) | 10 (10)
depression (Psychiatric disorders) | 17 (17) | 9 (10)
Mucositis/stomatitis (Gastrointestinal disorders) | 37 (37) | 9 (9)
Myalgias (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Musculoskeletal/Soft Tissue - other (Musculoskeletal and connective tissue disorders) | 13 (13) | 3 (4)
Nausea (Gastrointestinal disorders) | 64 (67) | 20 (20)
neuropathy (Nervous system disorders) | 47 (47) | 29 (29)
Neutropenia (Investigations) | 51 (63) | 17 (19)
Pain - abdomen (General disorders) | 3 (3) | 4 (5)
pain - back (Musculoskeletal and connective tissue disorders) | 13 (14) | 3 (3)
pain - breast (General disorders) | 9 (9) | 4 (4)
Pain - extremity (Musculoskeletal and connective tissue disorders) | 10 (10) | 11 (11)
Pain - headache (General disorders) | 17 (19) | 17 (18)
Pain - joint (Musculoskeletal and connective tissue disorders) | 7 (8) | 6 (6)
Pain chest (General disorders) | 5 (5) | 3 (3)
Pain - other (General disorders) | 17 (17) | 6 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 40 (44) | 3 (3)
Potassium serum high (Metabolism and nutrition disorders) | 5 (5) | 2 (2)
Potassium serum low (Metabolism and nutrition disorders) | 21 (21) | 5 (5)
Pruritus (itching) (Skin and subcutaneous tissue disorders) | 7 (7) | 3 (3)
Neurology - other (Nervous system disorders) | 13 (13) | 9 (9)
Desquamation (skin scaling) (Skin and subcutaneous tissue disorders) | 8 (8) | 2 (2)
Acne/acneiform (Skin and subcutaneous tissue disorders) | 19 (19) | 4 (4)
Hyponatremia (Metabolism and nutrition disorders) | 15 (15) | 11 (12)
dysgeusia (taste alteration) (Nervous system disorders) | 9 (10) | 14 (15)
hypothyroidism (Endocrine disorders) | 6 (6) | 3 (3)
Sexual/Reproduction -dryness, soreness, itching (Reproductive system and breast disorders) | 7 (7) | 2 (2)
Vomiting (Gastrointestinal disorders) | 13 (13) | 7 (9)
weight changes (gain or loss) (Investigations) | 6 (6) | 3 (3)
visual disorders - other (Eye disorders) | 10 (10) | 4 (4)
Fever (General disorders) | 6 (6) | 2 (2)
Gastrointestinal - Other (Gastrointestinal disorders) | 8 (8) | 2 (2)
Infection - upper respiratory (Infections and infestations) | 3 (3) | 5 (6)
Upper Respiratory - other (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 6 (6)
Renal/Genitourinary - Other (Renal and urinary disorders) | 6 (6) | 5 (5)
Auditory - other (Ear and labyrinth disorders) | 5 (5) | 2 (2)

LIMITATIONS AND CAVEATS:
The number of participants in each arm will not necessarily coincide with the number of participants affected in the respective arm. Some participants my have more than one event and/or some participants may not have an event at all.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days